CLINICAL TRIAL: NCT05200793
Title: A Comparative Clinical Study Evaluating the Efficacy of Empagliflozin or Linagliptin as an Alternative to Metformin for Treatment of Polycystic Ovary Syndrome in Egyptian Women
Brief Title: Efficacy of Empagliflozin or Linagliptin as an Alternative to Metformin for Treatment of Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Ibrahim ElMallah, Professor of Pharmacology & Therapeutics, Faculty of Pharmacy, Alexandria University, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201566
Record Dates: First submitted 2021-12-12; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: PCOS; Empagliflozin; Linagliptin; Metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — empagliflozin; Linagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metformin arm (control group) (Active Comparator): Patients will receive Metformin (1500 mg orally/day) for 12 weeks .
  Interventions: Drug: Metformin 1500 mg
- Empagliflozin arm (Active Comparator): Patients will receive Empagliflozin (25 mg orally/day) for 12 weeks.
  Interventions: Drug: Empagliflozin 25 mg
- Linagliptin arm (Active Comparator): Patients will receive Linagliptin (10 mg orally/day) for 12 weeks
  Interventions: Drug: Linagliptin 10 mg

INTERVENTIONS:
Drug: Empagliflozin 25 mg — This study is to compare the efficacy of Empagliflozin or Linagliptin as an alternative to Metformin for treatment of non-diabetic patients with polycystic ovary syndrome (PCOS)
  Other Names: Empagliflozin
  Arms: Empagliflozin arm
Drug: Linagliptin 10 mg — This study is to compare the efficacy of Empagliflozin or Linagliptin as an alternative to Metformin for treatment of non-diabetic patients with polycystic ovary syndrome (PCOS)
  Other Names: Linagliptin
  Arms: Linagliptin arm
Drug: Metformin 1500 mg — This study is to compare the efficacy of Empagliflozin or Linagliptin as an alternative to Metformin for treatment of non-diabetic patients with polycystic ovary syndrome (PCOS)
  Other Names: Metformin
  Arms: Metformin arm (control group)

SUMMARY:
The study aims to compare the efficacy of Empagliflozin or Linagliptin as an alternative to Metformin for treatment of non-diabetic patients with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
Patients with polycystic ovary syndrome will be randomized to three arms:

* Metformin (standard care)
* Empagliflozin or Linagliptin Resolution of the syndrome in addition to normalization of sex hormones, metabolic and inflammatory parameters will be tested

ELIGIBILITY:
Inclusion Criteria:

1. Women diagnosed with PCOS according to National Institute of Health criteria.
2. Age: >18 <40 years.
3. Infertile women (primary or secondary infertility).

Exclusion Criteria:

1. Patients with history of diabetes mellitus (Type 1 or 2).
2. Patients with liver or renal dysfunction; inflammatory diseases; autoimmune disease; cancer, acute cardiovascular event within last three months and uncontrolled endocrine or metabolic disease.
3. Significantly elevated triglyceride levels (fasting triglyceride > 400 mg/dL)
4. Untreated or poorly controlled hypertension (sitting blood pressure > 160/95 mm Hg).
5. Use of hormonal medications, lipid-lowering (statins, etc.), anti-obesity drugs or weight loss medications (prescription or OTC) and medications known to exacerbate glucose tolerance (such as isotretinoin, hormonal contraceptives, glucocorticoids, anabolic steroids) stopped for at least 8 weeks. Use of anti-androgens that act peripherally to reduce hirsutism such as 5-alpha reductase inhibitors stopped for at least 4 weeks.
6. Patients at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should have careful monitoring of their volume status.
7. Presence of hypersensitivity to Empagliflozin or other Sodium/glucose cotransporter 2 (SGLT2) inhibitors (e.g. anaphylaxis, angioedema, exfoliative skin conditions).
8. Known hypersensitivity or contraindications to use dipeptidyl peptidase-4 (DPP-4) inhibitors (saxagliptin, linagliptin, sitagliptin…).
9. Use of Metformin, Thiazolidinediones, glucagon-like peptide-1 (GLP-1) receptor agonists, DPP-4 inhibitors, SGLT2 inhibitors stopped for at least 4 weeks.
10. Eating disorders (anorexia, bulimia) or gastrointestinal disorders.
11. Having a history of bariatric surgery.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is for the treatment of polycystic ovary syndrome (PCOS)
Enrollment: 75 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Fertility parameters | 3-6 months
  [luteinizing hormone (LH)
Follicle-stimulating hormone | 3-6 months
  FSH
Free androgen index | 3-6 months
  total testosterone & sex hormone binding globulin (SHBG)
Transvaginal ultrasonography | 3-6 months
  disappearance of PCOS
Menstrual diaries | 3-6 months
  regulate menses cycles

SECONDARY OUTCOMES:
Metabolic parameters | 3-6 months
  Fasting blood glucose level
Lipid profile (metabolic parameters) | 3-6 months
  Total cholesterol, Low density lipoprotein (LDL), very low density lipoprotein (VLDL), high density lipoprotein (HDL), triglycerides (TG), atherogenic index I, II
Inflammatory indices | 3-6 months
  Interleukin 6 or Toll Like receptor 2

CONTACTS AND LOCATIONS:
Overall Officials: Hanan N Abdel Hafez, PhD, Study Chair — Professor of Obstetrics and Gynecology, Faculty of Medicine Mansoura University; Ahmed I ElMallah, PhD, Principal Investigator — Professor of Pharmacology and Therapeutics, Faculty of Pharmacy Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt